CLINICAL TRIAL: NCT04868188
Title: An Observational Pharmacokinetic Study of Intravenous Voriconazole Used for Treatment of Invasive Aspergillosis in Adult Patients With Severe Influenza / COVID-19 Supported With Extra-corporeal Membrane Oxygenation (ECMO)
Brief Title: Pharmacokinetics of Voriconazole in Adult ECMO Patients
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 136965 V1.0
Record Dates: First submitted 2021-02-18; First posted 2021-04-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Aspergillosis; Influenza; Covid19
Keywords: Voriconazole; Extracorporeal Membrane Oxygenation
MeSH Terms: conditions — Aspergillosis; Influenza, Human; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Voriconazole administration to adult patients with suspected fungal disease, receiving ECMO support: Adult (>18 years) patients with severe influenza / Covid-19 supported on ECMO and with confirmed or suspected aspergillosis infection.
  Interventions: Other: 5 blood samples; Genetic: Determination of CYP2C19 genotype

INTERVENTIONS:
Other: 5 blood samples — 5 blood samples across 3 occasions/sampling windows (Day 1-4, Day 6-9 and Day 11-14) to determine plasma concentrations of voriconazole
Genetic: Determination of CYP2C19 genotype — A single buccal swab to determine the CYP2C19 genotype will be undertaken during the course of ICU stay.

SUMMARY:
Given the high burden of fungal co-infection in patients admitted to ICU and improved outcomes with prompt anti-fungal treatment, it is of vital importance that the doses of anti-fungal are optimum to improve the dismal outcome of influenza/Covid-19 Associated Pulmonary Aspergillosis.

Due to the reported difficulties in dosing appropriately in ECMO patients, a prospective observational study is required to accurately evaluate the pharmacokinetics of voriconazole in patients supported on ECMO. This is to ensure that the dose of voriconazole is optimised to improve efficacy and reduce toxicity.

DETAILED DESCRIPTION:
A single centre, open label, prospective, observational, pharmacokinetic study of voriconazole administered to adults (aged > 18 years) supported on ECMO. This is a low-interventional study. There will be no treatment changes as a result of participation in this study. The decision to initiate voriconazole therapy will be taken independent of this study protocol. Intravenous voriconazole will be prescribed according to the approved dose in the SmPC. All adults requiring voriconazole therapy will be eligible for recruitment into the study.

The only additional procedure in this study will be to take a total of 5 blood samples across 3 occasions/sampling windows (Day 1-4, Day 6-9 and Day 11-14) to determine plasma concentrations of voriconazole. In addition, a single buccal swab to determine the CYP2C19 genotype will be undertaken during the course of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years
2. Admitted to ICU on ECMO support
3. Positive influenza or SARS-CoV-2 PCR from nasal, throat swab, BAL or other respiratory specimen.
4. Positive invasive aspergillosis infection (positive Aspergillus species culture from respiratory specimen or positive serum galactomannan) or strong clinical suspicion of invasive aspergillosis infection based on symptoms, CT, CXR.

Exclusion Criteria:

1. No participants < 18 years of age
2. Not requiring ECMO support
3. No positive influenza or SARS-CoV-2 results
4. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with acute (cardio-)respiratory failure, inadequately supported by mechanical ventilation, requiring additional support with ECMO, and in the opinion of the direct care team requires intravenous voriconazole therapy for treatment of confirmed or suspected invasive aspergillosis, will be eligible to be recruited.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Plasma levels of voriconazole administered to critically ill adult patients with suspected fungal disease, receiving ECMO support. | 14 days
  Primary parameter: Clearance (CL)
Plasma levels of voriconazole administered to critically ill adult patients with suspected fungal disease, receiving ECMO support. | 14 days
  Primary parameter: Volume of distribution (V)
Plasma levels of voriconazole administered to critically ill adult patients with suspected fungal disease, receiving ECMO support. | 14 days
  Secondary parameters: Maximum plasma concentration (Cmax)
Plasma levels of voriconazole administered to critically ill adult patients with suspected fungal disease, receiving ECMO support. | 14 days
  Secondary parameters: Area under plasma concentration time curve (AUC)
Plasma levels of voriconazole administered to critically ill adult patients with suspected fungal disease, receiving ECMO support. | 14 days
  Secondary parameters: Half-life (t1/2)

SECONDARY OUTCOMES:
To assess the influence of CYP2C19 genotype on the plasma levels of voriconazole | 14 days
  CYP2C19 genotype: identify *2, *3, and *17 mutations and any influence on plasma levels of voriconazole

CONTACTS AND LOCATIONS:
Overall Officials: Hakeem Yusuff, MD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No